CLINICAL TRIAL: NCT03843957
Title: Effectiveness and Implementation of mPATH-CRC: a Mobile Health System for Colorectal Cancer Screening
Brief Title: Effectiveness and Implementation of mPATH-CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00048919; R01CA218416 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Cancer; Rectum Cancer; Colon Cancer
Keywords: Mortality; Cancer Screening; Cancer Intervention; Mobile Health; Implementation Science
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Post-Implementation) (Experimental): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-CRC; Other: mPATH-Checkin; Other: "high touch" Implementation strategy
- Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Post-Implementation) (Experimental): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-CRC; Other: mPATH-Checkin; Other: "low touch" Implementation Strategy
- Clinic personnel on "high touch" Strategy (Post-Implementation) (Experimental): Clinic personnel (e.g., administrators, nurses, providers) who are involved with the implementation of mPATH-CRC, in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-CRC; Other: mPATH-Checkin; Other: "high touch" Implementation strategy
- Clinic personnel on "low touch" Strategy (Post-Implementation) (Experimental): Clinic personnel (e.g., administrators, nurses, providers) who are involved with the implementation of mPATH-CRC, in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-CRC; Other: mPATH-Checkin; Other: "low touch" Implementation Strategy
- All Adult Clinic Patients on "high touch" Strategy (Post-Implementation) (Experimental): English or Spanish-speaking patients aged 18 or older who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-Checkin; Other: "high touch" Implementation strategy
- All Adult Clinic Patients on "low touch" Strategy (Post-Implementation) (Experimental): English or Spanish-speaking patients aged 18 or older who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  Interventions: Other: mPATH-Checkin; Other: "low touch" Implementation Strategy
- Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Pre-Implementation) (Other): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy but in 8 months before implementation.
  Interventions: Other: "high touch" Implementation strategy
- Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Pre-Implementation) (Other): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy but in 8 months before implementation.
  Interventions: Other: "low touch" Implementation Strategy

INTERVENTIONS:
Other: mPATH-CRC — mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  Arms: Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Post-Implementation); Clinic personnel on "high touch" Strategy (Post-Implementation); Clinic personnel on "low touch" Strategy (Post-Implementation)
Other: mPATH-Checkin — The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  Arms: All Adult Clinic Patients on "high touch" Strategy (Post-Implementation); All Adult Clinic Patients on "low touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Post-Implementation); Clinic personnel on "high touch" Strategy (Post-Implementation); Clinic personnel on "low touch" Strategy (Post-Implementation)
Other: "high touch" Implementation strategy — The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
  Arms: All Adult Clinic Patients on "high touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "high touch" Strategy (Pre-Implementation); Clinic personnel on "high touch" Strategy (Post-Implementation)
Other: "low touch" Implementation Strategy — Clinics randomized to receive the low touch implementation strategy will receive:
  Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
  Arms: All Adult Clinic Patients on "low touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Post-Implementation); Clinic Patients Eligible for CRC Screening on "low touch" Strategy (Pre-Implementation); Clinic personnel on "low touch" Strategy (Post-Implementation)

SUMMARY:
Study Investigators are conducting this study to learn how to best implement a new iPad program in clinical practice.

DETAILED DESCRIPTION:
The study team has developed mPATH-CRC (mobile PAtient Technology for Health-Colorectal Cancer), a patient-friendly iPad program used by individuals immediately before a routine primary care visit. mPATH-CheckIn is a module that is used in conjunction with mPATH-CRC that consists of questions asked of all adult patients at check-in. mPATH-CRC is a module specific for patients due for CRC screening.

To fully realize mPATH-CRC's potential to decrease CRC mortality, the program now must be implemented in primary care practices in a way that encourages routine and sustained use. However, while hundreds of mobile health (mHealth) tools have been developed in recent years, the optimal strategies for implementing and maintaining mHealth interventions in clinical practice are unknown. This study will compare the results of a "high touch" strategy to a "low touch" strategy using a Type III hybrid design and incorporating mixed methods to evaluate implementation, maintenance, and effectiveness of mPATH-CRC in a diverse sample of community-based practices.

The study will be conducted in three phases: 1) in a cluster-randomized controlled trial of 22 primary care clinics, the study team will compare the implementation outcomes of a "high touch" evidence-based mHealth implementation strategy with a "low touch" implementation strategy; 2) in a nested pragmatic study, the study team will estimate the effect of mPATH-CRC on completion of CRC screening within 16 weeks of a clinic visit; and 3) by surveying and interviewing clinic staff and providers after implementation is complete, the study team will determine the factors that facilitate or impede the maintenance of mHealth interventions.

ELIGIBILITY:
This study will include three distinct populations of participants: 1) healthcare providers and staff at primary care practices, 2) patients aged 18 and older seen in the participating study sites, and 3) patients aged 50-74 seen in the participating study sites who are eligible for CRC screening

Patient Inclusion Criteria:

Due for routine CRC screening, defined as:

* No colonoscopy within the prior 10 years
* No flexible sigmoidoscopy within the prior 5 years
* No CT colonography within the prior 5 years
* No fecal DNA testing within the prior 3 years
* No fecal blood testing (guaiac-based test with home kit or fecal immunochemical test) within the prior 12 months

Patient Exclusion Criteria:

* Personal history of CRC
* First degree relative with CRC
* Personal history of colorectal polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77145 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified participant data that underlie the results reported in peer-reviewed publications (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Investigators who provide a methodologically sound proposal to use the participant data in a meta-analysis.

REFERENCES:
- [Background] Sharp L, Tilson L, Whyte S, O'Ceilleachair A, Walsh C, Usher C, Tappenden P, Chilcott J, Staines A, Barry M, Comber H. Cost-effectiveness of population-based screening for colorectal cancer: a comparison of guaiac-based faecal occult blood testing, faecal immunochemical testing and flexible sigmoidoscopy. Br J Cancer. 2012 Feb 28;106(5):805-16. doi: 10.1038/bjc.2011.580. Epub 2012 Feb 16. PMID 22343624
- [Background] Lin JS, Piper MA, Perdue LA, Rutter CM, Webber EM, O'Connor E, Smith N, Whitlock EP. Screening for Colorectal Cancer: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2016 Jun 21;315(23):2576-94. doi: 10.1001/jama.2016.3332. PMID 27305422
- [Background] Knudsen AB, Zauber AG, Rutter CM, Naber SK, Doria-Rose VP, Pabiniak C, Johanson C, Fischer SE, Lansdorp-Vogelaar I, Kuntz KM. Estimation of Benefits, Burden, and Harms of Colorectal Cancer Screening Strategies: Modeling Study for the US Preventive Services Task Force. JAMA. 2016 Jun 21;315(23):2595-609. doi: 10.1001/jama.2016.6828. PMID 27305518
- [Background] Inadomi JM. Screening for Colorectal Neoplasia. N Engl J Med. 2017 Jan 12;376(2):149-156. doi: 10.1056/NEJMcp1512286. No abstract available. PMID 28076720
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FAR, Gillman MW, Harper DM, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Owens DK, Phillips WR, Phipps MG, Pignone MP, Siu AL. Screening for Colorectal Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jun 21;315(23):2564-2575. doi: 10.1001/jama.2016.5989. PMID 27304597
- [Background] Qaseem A, Denberg TD, Hopkins RH Jr, Humphrey LL, Levine J, Sweet DE, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Screening for colorectal cancer: a guidance statement from the American College of Physicians. Ann Intern Med. 2012 Mar 6;156(5):378-86. doi: 10.7326/0003-4819-156-5-201203060-00010. PMID 22393133
- [Background] Smith RA, Andrews K, Brooks D, DeSantis CE, Fedewa SA, Lortet-Tieulent J, Manassaram-Baptiste D, Brawley OW, Wender RC. Cancer screening in the United States, 2016: A review of current American Cancer Society guidelines and current issues in cancer screening. CA Cancer J Clin. 2016 Mar-Apr;66(2):96-114. doi: 10.3322/caac.21336. Epub 2016 Jan 21. PMID 26797525
- [Background] Rex DK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Levin TR, Lieberman D, Robertson DJ. Colorectal Cancer Screening: Recommendations for Physicians and Patients from the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2017 Jul;112(7):1016-1030. doi: 10.1038/ajg.2017.174. Epub 2017 Jun 6. PMID 28555630
- [Background] White A, Thompson TD, White MC, Sabatino SA, de Moor J, Doria-Rose PV, Geiger AM, Richardson LC. Cancer Screening Test Use - United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 3;66(8):201-206. doi: 10.15585/mmwr.mm6608a1. PMID 28253225
- [Background] Gupta S, Sussman DA, Doubeni CA, Anderson DS, Day L, Deshpande AR, Elmunzer BJ, Laiyemo AO, Mendez J, Somsouk M, Allison J, Bhuket T, Geng Z, Green BB, Itzkowitz SH, Martinez ME. Challenges and possible solutions to colorectal cancer screening for the underserved. J Natl Cancer Inst. 2014 Apr;106(4):dju032. doi: 10.1093/jnci/dju032. Epub 2014 Mar 28. PMID 24681602
- [Background] Yao N, Alcala HE, Anderson R, Balkrishnan R. Cancer Disparities in Rural Appalachia: Incidence, Early Detection, and Survivorship. J Rural Health. 2017 Sep;33(4):375-381. doi: 10.1111/jrh.12213. Epub 2016 Sep 7. PMID 27602545
- [Background] Doubeni CA, Laiyemo AO, Major JM, Schootman M, Lian M, Park Y, Graubard BI, Hollenbeck AR, Sinha R. Socioeconomic status and the risk of colorectal cancer: an analysis of more than a half million adults in the National Institutes of Health-AARP Diet and Health Study. Cancer. 2012 Jul 15;118(14):3636-44. doi: 10.1002/cncr.26677. Epub 2012 Jan 3. PMID 22898918
- [Background] James TM, Greiner KA, Ellerbeck EF, Feng C, Ahluwalia JS. Disparities in colorectal cancer screening: a guideline-based analysis of adherence. Ethn Dis. 2006 Winter;16(1):228-33. PMID 16599375
- [Background] Morgan JW, Cho MM, Guenzi CD, Jackson C, Mathur A, Natto Z, Kazanjian K, Tran H, Shavlik D, Lum SS. Predictors of delayed-stage colorectal cancer: are we neglecting critical demographic information? Ann Epidemiol. 2011 Dec;21(12):914-21. doi: 10.1016/j.annepidem.2011.09.002. Epub 2011 Oct 13. PMID 22000327
- [Background] Siegel R, Desantis C, Jemal A. Colorectal cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):104-17. doi: 10.3322/caac.21220. Epub 2014 Mar 17. PMID 24639052
- [Background] Miller DP Jr, Brownlee CD, McCoy TP, Pignone MP. The effect of health literacy on knowledge and receipt of colorectal cancer screening: a survey study. BMC Fam Pract. 2007 Mar 30;8:16. doi: 10.1186/1471-2296-8-16. PMID 17394668
- [Background] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Oldach BR, Katz ML. Health literacy and cancer screening: a systematic review. Patient Educ Couns. 2014 Feb;94(2):149-57. doi: 10.1016/j.pec.2013.10.001. Epub 2013 Oct 14. PMID 24207115
- [Background] Beydoun HA, Beydoun MA. Predictors of colorectal cancer screening behaviors among average-risk older adults in the United States. Cancer Causes Control. 2008 May;19(4):339-59. doi: 10.1007/s10552-007-9100-y. Epub 2007 Dec 18. PMID 18085415
- [Background] Weinberg DS, Turner BJ, Wang H, Myers RE, Miller S. A survey of women regarding factors affecting colorectal cancer screening compliance. Prev Med. 2004 Jun;38(6):669-75. doi: 10.1016/j.ypmed.2004.02.015. PMID 15193887
- [Background] Berkowitz Z, Hawkins NA, Peipins LA, White MC, Nadel MR. Beliefs, risk perceptions, and gaps in knowledge as barriers to colorectal cancer screening in older adults. J Am Geriatr Soc. 2008 Feb;56(2):307-14. doi: 10.1111/j.1532-5415.2007.01547.x. Epub 2007 Dec 7. PMID 18070002
- [Background] Farmer MM, Bastani R, Kwan L, Belman M, Ganz PA. Predictors of colorectal cancer screening from patients enrolled in a managed care health plan. Cancer. 2008 Mar 15;112(6):1230-8. doi: 10.1002/cncr.23290. PMID 18266204
- [Background] Wee CC, McCarthy EP, Phillips RS. Factors associated with colon cancer screening: the role of patient factors and physician counseling. Prev Med. 2005 Jul;41(1):23-9. doi: 10.1016/j.ypmed.2004.11.004. Epub 2004 Dec 29. PMID 15916989
- [Background] Klabunde CN, Schenck AP, Davis WW. Barriers to colorectal cancer screening among Medicare consumers. Am J Prev Med. 2006 Apr;30(4):313-9. doi: 10.1016/j.amepre.2005.11.006. PMID 16530618
- [Background] Seeff LC, Nadel MR, Klabunde CN, Thompson T, Shapiro JA, Vernon SW, Coates RJ. Patterns and predictors of colorectal cancer test use in the adult U.S. population. Cancer. 2004 May 15;100(10):2093-103. doi: 10.1002/cncr.20276. PMID 15139050
- [Background] Ayres CG, Griffith HM. Perceived barriers to and facilitators of the implementation of priority clinical preventive services guidelines. Am J Manag Care. 2007 Mar;13(3):150-5. PMID 17335358
- [Background] Yarnall KS, Pollak KI, Ostbye T, Krause KM, Michener JL. Primary care: is there enough time for prevention? Am J Public Health. 2003 Apr;93(4):635-41. doi: 10.2105/ajph.93.4.635. PMID 12660210
- [Background] Ostbye T, Yarnall KS, Krause KM, Pollak KI, Gradison M, Michener JL. Is there time for management of patients with chronic diseases in primary care? Ann Fam Med. 2005 May-Jun;3(3):209-14. doi: 10.1370/afm.310. PMID 15928223
- [Background] Katz ML, Broder-Oldach B, Fisher JL, King J, Eubanks K, Fleming K, Paskett ED. Patient-provider discussions about colorectal cancer screening: who initiates elements of informed decision making? J Gen Intern Med. 2012 Sep;27(9):1135-41. doi: 10.1007/s11606-012-2045-1. Epub 2012 Apr 5. PMID 22476985
- [Background] Zapka JM, Klabunde CN, Arora NK, Yuan G, Smith JL, Kobrin SC. Physicians' colorectal cancer screening discussion and recommendation patterns. Cancer Epidemiol Biomarkers Prev. 2011 Mar;20(3):509-21. doi: 10.1158/1055-9965.EPI-10-0749. Epub 2011 Jan 14. PMID 21239688
- [Background] Anhang Price R, Zapka J, Edwards H, Taplin SH. Organizational factors and the cancer screening process. J Natl Cancer Inst Monogr. 2010;2010(40):38-57. doi: 10.1093/jncimonographs/lgq008. PMID 20386053
- [Background] Taplin SH, Anhang Price R, Edwards HM, Foster MK, Breslau ES, Chollette V, Prabhu Das I, Clauser SB, Fennell ML, Zapka J. Introduction: Understanding and influencing multilevel factors across the cancer care continuum. J Natl Cancer Inst Monogr. 2012 May;2012(44):2-10. doi: 10.1093/jncimonographs/lgs008. PMID 22623590
- [Background] Miller DP Jr, Weaver KE, Case LD, Babcock D, Lawler D, Denizard-Thompson N, Pignone MP, Spangler JG. Usability of a Novel Mobile Health iPad App by Vulnerable Populations. JMIR Mhealth Uhealth. 2017 Apr 11;5(4):e43. doi: 10.2196/mhealth.7268. PMID 28400354
- [Background] Orr JA, King RJ. Mobile phone SMS messages can enhance healthy behaviour: a meta-analysis of randomised controlled trials. Health Psychol Rev. 2015;9(4):397-416. doi: 10.1080/17437199.2015.1022847. Epub 2015 May 28. PMID 25739668
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Ostrander RE, Thompson HJ, Demiris G. Using targeted messaging to increase physical activity in older adults: a review. J Gerontol Nurs. 2014 Sep;40(9):36-48. doi: 10.3928/00989134-20140324-03. Epub 2014 Mar 31. PMID 24694043
- [Background] Vodopivec-Jamsek V, de Jongh T, Gurol-Urganci I, Atun R, Car J. Mobile phone messaging for preventive health care. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007457. doi: 10.1002/14651858.CD007457.pub2. PMID 23235643
- [Background] Hawley S, Lillie S, Cooper G, Elston Lafata J. Managed care patients' preferences, physician recommendations, and colon cancer screening. Am J Manag Care. 2014 Jul;20(7):555-61. PMID 25295401
- [Background] Inadomi JM, Vijan S, Janz NK, Fagerlin A, Thomas JP, Lin YV, Munoz R, Lau C, Somsouk M, El-Nachef N, Hayward RA. Adherence to colorectal cancer screening: a randomized clinical trial of competing strategies. Arch Intern Med. 2012 Apr 9;172(7):575-82. doi: 10.1001/archinternmed.2012.332. PMID 22493463
- [Background] Miller DP Jr, Spangler JG, Case LD, Goff DC Jr, Singh S, Pignone MP. Effectiveness of a web-based colorectal cancer screening patient decision aid: a randomized controlled trial in a mixed-literacy population. Am J Prev Med. 2011 Jun;40(6):608-15. doi: 10.1016/j.amepre.2011.02.019. PMID 21565651
- [Background] Miller DP, Denizard-Thompson N, Case LD, Weaver KE, Pignone MP, Lawler D, Troyer J, Spangler JG. The effect of a mobile health intervention (mPATH-CRC) on colorectal cancer screening in a diverse patient population. J Gen Intern Med. 2017 Apr;32(2 Supplement):S338
- [Background] Sabatino SA, White MC, Thompson TD, Klabunde CN; Centers for Disease Control and Prevention (CDC). Cancer screening test use - United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 May 8;64(17):464-8. PMID 25950253
- [Background] Bardus M, Smith JR, Samaha L, Abraham C. Mobile Phone and Web 2.0 Technologies for Weight Management: A Systematic Scoping Review. J Med Internet Res. 2015 Nov 16;17(11):e259. doi: 10.2196/jmir.5129. PMID 26573984
- [Background] Matthew-Maich N, Harris L, Ploeg J, Markle-Reid M, Valaitis R, Ibrahim S, Gafni A, Isaacs S. Designing, Implementing, and Evaluating Mobile Health Technologies for Managing Chronic Conditions in Older Adults: A Scoping Review. JMIR Mhealth Uhealth. 2016 Jun 9;4(2):e29. doi: 10.2196/mhealth.5127. PMID 27282195
- [Background] Joe J, Demiris G. Older adults and mobile phones for health: a review. J Biomed Inform. 2013 Oct;46(5):947-54. doi: 10.1016/j.jbi.2013.06.008. Epub 2013 Jun 25. PMID 23810858
- [Background] Bandura A. Social Foundations of Thought and Action: A Social Cognitive Theory. 1 edition. Englewood Cliffs, N.J: Prentice Hall; 1985
- [Background] Weaver KE, Ellis SD, Denizard-Thompson N, Kronner D, Miller DP. Crafting Appealing Text Messages to Encourage Colorectal Cancer Screening Test Completion: A Qualitative Study. JMIR Mhealth Uhealth. 2015 Nov 4;3(4):e100. doi: 10.2196/mhealth.4651. PMID 26537553
- [Background] Seale JP, Johnson JA, Clark DC, Shellenberger S, Pusser AT, Dhabliwala J, Sigman EJ, Dittmer T, Barnes Le K, Miller DP, Clemow D. A Multisite Initiative to Increase the Use of Alcohol Screening and Brief Intervention Through Resident Training and Clinic Systems Changes. Acad Med. 2015 Dec;90(12):1707-12. doi: 10.1097/ACM.0000000000000846. PMID 26200578
- [Background] Venkatesh V, Bala H. Technology Acceptance Model 3 and a Research Agenda on Interventions. Decis Sci. 2008 May 1;39(2):273-315.
- [Background] Venkatesh V, Davis FD. A Theoretical Extension of the Technology Acceptance Model: Four Longitudinal Field Studies. Manag Sci. 2000 Feb;46(2):186-204.
- [Background] Chan WV, Pearson TA, Bennett GC, Cushman WC, Gaziano TA, Gorman PN, Handler J, Krumholz HM, Kushner RF, MacKenzie TD, Sacco RL, Smith SC Jr, Stevens VJ, Wells BL. ACC/AHA Special Report: Clinical Practice Guideline Implementation Strategies: A Summary of Systematic Reviews by the NHLBI Implementation Science Work Group: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Feb 28;69(8):1076-1092. doi: 10.1016/j.jacc.2016.11.004. Epub 2017 Jan 26. PMID 28132746
- [Background] Ivers NM, Sales A, Colquhoun H, Michie S, Foy R, Francis JJ, Grimshaw JM. No more 'business as usual' with audit and feedback interventions: towards an agenda for a reinvigorated intervention. Implement Sci. 2014 Jan 17;9:14. doi: 10.1186/1748-5908-9-14. PMID 24438584
- [Background] Ford JH 2nd, Alagoz E, Dinauer S, Johnson KA, Pe-Romashko K, Gustafson DH. Successful Organizational Strategies to Sustain Use of A-CHESS: A Mobile Intervention for Individuals With Alcohol Use Disorders. J Med Internet Res. 2015 Aug 18;17(8):e201. doi: 10.2196/jmir.3965. PMID 26286257
- [Background] Stetler CB, Legro MW, Wallace CM, Bowman C, Guihan M, Hagedorn H, Kimmel B, Sharp ND, Smith JL. The role of formative evaluation in implementation research and the QUERI experience. J Gen Intern Med. 2006 Feb;21 Suppl 2(Suppl 2):S1-8. doi: 10.1111/j.1525-1497.2006.00355.x. PMID 16637954
- [Background] Green LW, Glasgow RE. Evaluating the relevance, generalization, and applicability of research: issues in external validation and translation methodology. Eval Health Prof. 2006 Mar;29(1):126-53. doi: 10.1177/0163278705284445. PMID 16510882
- [Background] Shaw EK, Howard J, West DR, Crabtree BF, Nease DE Jr, Tutt B, Nutting PA. The role of the champion in primary care change efforts: from the State Networks of Colorado Ambulatory Practices and Partners (SNOCAP). J Am Board Fam Med. 2012 Sep-Oct;25(5):676-85. doi: 10.3122/jabfm.2012.05.110281. PMID 22956703
- [Background] Chambers DA, Glasgow RE, Stange KC. The dynamic sustainability framework: addressing the paradox of sustainment amid ongoing change. Implement Sci. 2013 Oct 2;8:117. doi: 10.1186/1748-5908-8-117. PMID 24088228
- [Background] Neta G, Glasgow RE, Carpenter CR, Grimshaw JM, Rabin BA, Fernandez ME, Brownson RC. A Framework for Enhancing the Value of Research for Dissemination and Implementation. Am J Public Health. 2015 Jan;105(1):49-57. doi: 10.2105/AJPH.2014.302206. PMID 25393182
- [Background] ATLAS.ti. Berlin: Scientific Software Development; 2013.
- [Background] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530
- [Background] Rutterford C, Copas A, Eldridge S. Methods for sample size determination in cluster randomized trials. Int J Epidemiol. 2015 Jun;44(3):1051-67. doi: 10.1093/ije/dyv113. Epub 2015 Jul 13. PMID 26174515
- [Background] Murray DM, Varnell SP, Blitstein JL. Design and analysis of group-randomized trials: a review of recent methodological developments. Am J Public Health. 2004 Mar;94(3):423-32. doi: 10.2105/ajph.94.3.423. PMID 14998806
- [Background] Austin PC. A comparison of the statistical power of different methods for the analysis of cluster randomization trials with binary outcomes. Stat Med. 2007 Aug 30;26(19):3550-65. doi: 10.1002/sim.2813. PMID 17238238
- [Background] Ma J, Thabane L, Kaczorowski J, Chambers L, Dolovich L, Karwalajtys T, Levitt C. Comparison of Bayesian and classical methods in the analysis of cluster randomized controlled trials with a binary outcome: the Community Hypertension Assessment Trial (CHAT). BMC Med Res Methodol. 2009 Jun 16;9:37. doi: 10.1186/1471-2288-9-37. PMID 19531226
- [Background] Wagner AK, Soumerai SB, Zhang F, Ross-Degnan D. Segmented regression analysis of interrupted time series studies in medication use research. J Clin Pharm Ther. 2002 Aug;27(4):299-309. doi: 10.1046/j.1365-2710.2002.00430.x. PMID 12174032
- [Background] Penfold RB, Zhang F. Use of interrupted time series analysis in evaluating health care quality improvements. Acad Pediatr. 2013 Nov-Dec;13(6 Suppl):S38-44. doi: 10.1016/j.acap.2013.08.002. PMID 24268083
- [Background] Helfrich CD, Li YF, Sharp ND, Sales AE. Organizational readiness to change assessment (ORCA): development of an instrument based on the Promoting Action on Research in Health Services (PARIHS) framework. Implement Sci. 2009 Jul 14;4:38. doi: 10.1186/1748-5908-4-38. PMID 19594942
- [Derived] Miller DP Jr, Snavely AC, Dharod A, Wright E, Randazzo A, Bundy R, Dignan M, Foley KL. High-Touch vs Low-Touch Strategy for Implementing a CRC Screening Digital Health Intervention: A Randomized Clinical Trial. JAMA Intern Med. 2025 Jul 1;185(7):788-795. doi: 10.1001/jamainternmed.2025.0779. PMID 40323625
- [Derived] Snavely AC, Foley K, Dharod A, Dignan M, Brower H, Wright E, Miller DP Jr. Effectiveness and implementation of mPATH-CRC: a mobile health system for colorectal cancer screening. Trials. 2023 Apr 14;24(1):274. doi: 10.1186/s13063-023-07273-5. PMID 37060023
- See also: Kutner M, Greenburg E, Jin Y, Paulsen C. The Health Literacy of America's Adults: Results from the 2003 National Assessment of Adult Literacy. NCES 2006-483. Natl Cent Educ Stat [Internet]. 2006 [cited 2015 Sep 23]; — http://eric.ed.gov/?id=ED493284
- See also: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Health Statistics. Summary Health Statistics: National Health Interview Survey, 2015 [Internet]. [cited 2017 Jun 16]. — https://ftp.cdc.gov/pub/Health_Statistics/NCHS/NHIS/SHS/2015_SHS_Table_A-18.pdf
- See also: Monegain B. Cerner still leads in EHR marketshare, though smaller vendors are making moves. Healthc IT News [Internet]. 2017 Apr 28 [cited 2017 Jun 22]; — http://www.healthcareitnews.com/news/cerner-still-leads-ehr-marketshare-though-smaller-vendors-are-making-moves
- See also: Berta W, Cranley L, Dearing JW, Dogherty EJ, Squires JE, Estabrooks CA. Why (we think) facilitation works: insights from organizational learning theory. Implement Sci [Internet]. 2015 Dec [cited 2017 May 8];10(1). — http://implementationscience.biomedcentral.com/articles/10.1186/s13012-015-0323-0
- See also: Maher L, Gustafson D, Evans A. Sustainability Model and Guide [Internet]. British National Health Service Modernization Agency; 2004 [cited 2017 Jun 9]. — http://www.qihub.scot.nhs.uk/media/162236/sustainability_model.pdf
- See also: Soo S, Baker WB and GR. Role of Champions in the Implementation of Patient Safety Practice Change. Healthc Q [Internet]. 2009 Aug 15 [cited 2017 May 8]; — http://www.longwoods.com/content/20979
- See also: Behavioral Risk Factor Surveillance System, 2015 Questionnaire [Internet]. Centers for Disease Control and Prevention (US); 2014 [cited 2016 Sep 30]. — http://www.cdc.gov/brfss/questionnaires/pdf-ques/2015-brfss-questionnaire-12-29-14.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 clinics were enrolled in the study. These clinics were randomized to the "high touch" or "low touch" implementation strategy. From these 18 clinics, 77145 total participants were enrolled. This includes 67134 adult patients (13092 of whom were eligible for CRC screening) seen in the clinics sometime during the 12 months after implementation, 514 clinic personnel involved in the implementation of mPATH, and 9497 patients in the pre-implementation cohort (8 months prior to implementation).
Pre-assignment Details: This is a pragmatic trial, with data being pulled from the electronic health record, so there is no loss to follow-up. A patient enters the dataset once at the time of their clinic visit; they are not actively followed over time but rather a retrospective data pull was conducted at the end of the study for relevant outcomes. The periods described under the description for "high touch" and "low touch" are at the clinic level, not the patient level.
Units Other Than Participants: Clinics
Groups:
- "High Touch" Strategy: Populations evaluated include: Patients Eligible for CRC Screening (Pre- and Post-Implementation), All Adult Patients (Post-Implementation), and Clinic Personnel (Post-Implementation) at clinics randomized to the "high touch" strategy.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "high touch" Implementation strategy: The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- "Low Touch" Strategy: Populations evaluated include: Patients Eligible for CRC Screening (Pre- and Post-Implementation), All Adult Patients (Post-Implementation), and Clinic Personnel (Post-Implementation) at clinics randomized to the "low touch" strategy.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
Period: Overall Study
Arm/Group | "High Touch" Strategy | "Low Touch" Strategy
Started | 49583; 10 Clinics | 27562; 8 Clinics
All Adult Clinic Patients Post-Implementation: 18 or Older | 43775; 10 Clinics | 23359; 8 Clinics
Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Aged 50-74 | 7933; 10 Clinics | 5159; 8 Clinics
Clinic Personnel Post-Implementation | 282; 10 Clinics | 232; 8 Clinics
Adult Clinic Patients Eligible for CRC Screening Pre-Implementation: Aged 50-74 | 5526; 10 Clinics | 3971; 8 Clinics
Completed | 49583; 10 Clinics | 27562; 8 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- All Adult Clinic Patients on "High Touch" Strategy (Post-Implementation): English or Spanish-speaking patients aged 18 or older who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "high touch" Implementation strategy: The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- All Adult Clinic Patients on "Low Touch" Strategy (Post-Implementation): English or Spanish-speaking patients aged 18 or older who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Clinic Personnel on "High Touch" Strategy (Post-Implementation): Clinic personnel (e.g., administrators, nurses, providers) who are involved with the implementation of mPATH-CRC, in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "high touch" Implementation strategy: The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Clinic Personnel on "Low Touch" Strategy (Post-Implementation): Clinic personnel (e.g., administrators, nurses, providers) who are involved with the implementation of mPATH-CRC, in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Pre-Implementation): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy but in 8 months before implementation.
  "high touch" Implementation strategy: The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Pre-Implementation): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy but in 8 months before implementation.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Total: Total of all reporting groups
Arm/Group | All Adult Clinic Patients on "High Touch" Strategy (Post-Implementation) | All Adult Clinic Patients on "Low Touch" Strategy (Post-Implementation) | Clinic Personnel on "High Touch" Strategy (Post-Implementation) | Clinic Personnel on "Low Touch" Strategy (Post-Implementation) | Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Pre-Implementation) | Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Pre-Implementation) | Total
Number analyzed (Participants) | 43775 | 23359 | 282 | 232 | 5526 | 3971 | 77145
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographics data are only available for clinic personnel who filled out a survey. "Adult Clinic Patients Eligible for CRC Screening Post-Implementation" is a subset of "All Adult Clinic Patients (Post-Implementation)." The subset is included here because the patients eligible for CRC screening is the analysis population for outcomes related to implementation of mPATH-CRC.
  years
    All Participants: number analyzed (Participants) | 43775 | 23359 | 126 | 78 | 5526 | 3971 | 76835
    All Participants | 55.0 (17.7) | 52.3 (17.8) | 37.0 (8.8) | 37.6 (8.4) | 59.5 (7.1) | 59.4 (6.9) | 54.7 (16.9)
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: number analyzed (Participants) | 7933 | 5159 | 0 | 0 | 0 | 0 | 13092
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation | 59.9 (7.2) | 59.6 (6.9) |  |  |  |  | 59.8 (7.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: "Adult Clinic Patients Eligible for CRC Screening Post-Implementation" is a subset of "All Adult Clinic Patients (Post-Implementation)." The subset is included here because the patients eligible for CRC screening is the analysis population for outcomes related to implementation of mPATH-CRC.
  Participants
    All Participants: Male | 17952 | 9828 | 20 | 11 | 2389 | 1783 | 31983
    All Participants: Female | 25823 | 13530 | 162 | 108 | 3137 | 2188 | 44948
    All Participants: Unknown | 0 | 1 | 100 | 113 | 0 | 0 | 214
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: number analyzed (Participants) | 7933 | 5159 | 0 | 0 | 0 | 0 | 13092
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Male | 3504 | 2376 |  |  |  |  | 5880
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Female | 4429 | 2782 |  |  |  |  | 7211
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Unknown | 0 | 1 |  |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: "Adult Clinic Patients Eligible for CRC Screening Post-Implementation" is a subset of "All Adult Clinic Patients (Post-Implementation)." The subset is included here because the patients eligible for CRC screening is the analysis population for outcomes related to implementation of mPATH-CRC.
  Participants
    All Participants: Hispanic or Latino | 2412 | 955 | 14 | 7 | 361 | 114 | 3863
    All Participants: Not Hispanic or Latino | 41035 | 22286 | 162 | 107 | 5112 | 3840 | 72542
    All Participants: Unknown or Not Reported | 328 | 118 | 106 | 118 | 53 | 17 | 740
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: number analyzed (Participants) | 7933 | 5159 | 0 | 0 | 0 | 0 | 13092
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Hispanic or Latino | 444 | 195 |  |  |  |  | 639
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Not Hispanic or Latino | 7419 | 4937 |  |  |  |  | 12356
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Unknown or Not Reported | 70 | 27 |  |  |  |  | 97
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: "Adult Clinic Patients Eligible for CRC Screening Post-Implementation" is a subset of "All Adult Clinic Patients (Post-Implementation)." The subset is included here because the patients eligible for CRC screening is the analysis population for outcomes related to implementation of mPATH-CRC.
  Participants
    All Participants: American Indian or Alaska Native | 319 | 128 | 1 | 2 | 55 | 22 | 527
    All Participants: Asian | 930 | 504 | 5 | 4 | 115 | 86 | 1644
    All Participants: Native Hawaiian or Other Pacific Islander | 46 | 35 | 0 | 0 | 13 | 4 | 98
    All Participants: Black or African American | 4490 | 3329 | 31 | 19 | 656 | 533 | 9058
    All Participants: White | 35542 | 18286 | 135 | 85 | 4346 | 3181 | 61575
    All Participants: More than one race | 0 | 0 | 2 | 1 | 0 | 0 | 3
    All Participants: Unknown or Not Reported | 2448 | 1077 | 108 | 121 | 341 | 145 | 4240
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: number analyzed (Participants) | 7933 | 5159 | 0 | 0 | 0 | 0 | 13092
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: American Indian or Alaska Native | 63 | 44 |  |  |  |  | 107
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Asian | 154 | 99 |  |  |  |  | 253
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Native Hawaiian or Other Pacific Islander | 12 | 6 |  |  |  |  | 18
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Black or African American | 860 | 704 |  |  |  |  | 1564
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: White | 6387 | 4093 |  |  |  |  | 10480
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: More than one race | 0 | 0 |  |  |  |  | 0
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Unknown or Not Reported | 457 | 213 |  |  |  |  | 670
Insurance [Count of Participants; unit: Participants] — Population: "Adult Clinic Patients Eligible for CRC Screening Post-Implementation" is a subset of "All Adult Clinic Patients (Post-Implementation)." The subset is included here because the patients eligible for CRC screening is the analysis population for outcomes related to implementation of mPATH-CRC.
  Participants
    All Participants: Commercial | 23666 | 13028 | 0 | 0 | 2922 | 2124 | 41740
    All Participants: Medicare | 14644 | 6893 | 0 | 0 | 1857 | 1293 | 24687
    All Participants: Medicaid | 1783 | 1587 | 0 | 0 | 141 | 113 | 3624
    All Participants: Other | 1374 | 722 | 0 | 0 | 222 | 128 | 2446
    All Participants: Uninsured | 2308 | 1129 | 0 | 0 | 384 | 313 | 4134
    All Participants: Unknown | 0 | 0 | 282 | 232 | 0 | 0 | 514
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: number analyzed (Participants) | 7933 | 5159 | 0 | 0 | 0 | 0 | 13092
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Commercial | 4414 | 2880 |  |  |  |  | 7294
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Medicare | 2627 | 1648 |  |  |  |  | 4275
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Medicaid | 216 | 203 |  |  |  |  | 419
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Other | 273 | 140 |  |  |  |  | 413
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Uninsured | 403 | 288 |  |  |  |  | 691
    Adult Clinic Patients Eligible for CRC Screening Post-Implementation: Unknown | 0 | 0 |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Complete the mPATH-CRC Program
Description: mPATH-CRC Implementation: Percent of all eligible patients, ages 50 - 74, who complete the mPATH-CRC program in the 6th month following the implementation date.
Time Frame: Month 6
Population: The analysis population for this outcome is in the sixth month after implementation, so this is a subset of the overall baseline population that includes patients eligible for CRC screening over the full12 months following implementation.
Measure: Count of Participants; unit: Participants
Groups:
- Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Post-Implementation): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "high touch" Implementation strategy: The "high touch" strategy consists of pre-implementation activities, training, and ongoing support.
  Pre-Implementation Activities
  * Clinic champion identified.
  * Study team meeting with clinic champion
  * Implementation adaptations as needed for clinic flow
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  * Monthly program usage report sent to clinic champions
  * Scheduled phone-calls with clinic champion to review QA data and explore potential barriers.
  * Implementation adaptations as needed for clinic flow
  * Goal-triggered follow-up on-site trainings
  * Additional on-site trainings as requested.
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
- Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Post-Implementation): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "high touch" implementation strategy in the 12 months after implementation.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
Arm/Group | Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Post-Implementation) | Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Post-Implementation)
Number analyzed (Participants) | 558 | 397
Participants | 5 | 4

2. Secondary Outcome: mPATH-CRC Reach (by Socioeconomic Strata)
Description: mPATH-CRC Reach: The proportion of patients, ages 50 - 74, who are given mPATH-CRC or have risk factors identified by mPATH-CheckIn in months 1-6 by varying socioeconomic strata (Describe strata)
Time Frame: up to month 6
Reporting Status: Not Posted

3. Secondary Outcome: mPATH-CRC Adoption
Description: The mean usage of mPATH-CRC among staff and providers over the first 6 months following implementation; usage is calculated for each staff/provider as the proportion of times mPATH-CRC is completed out of the total times mPATH-CRC should have been launched.
Time Frame: up to month 6
Reporting Status: Not Posted

4. Secondary Outcome: mPATH-CheckIn Reach
Description: The proportion of patients aged 18 or older who complete mPATH-CheckIn in months 1-6; this outcome will be calculated overall and within socioeconomic strata
Time Frame: up to month 6
Reporting Status: Not Posted

5. Secondary Outcome: mPATH-CheckIn Adoption
Description: The mean usage of mPATH-CheckIn among staff and providers over the first 6 months following implementation; usage is calculated for front desk staff as the proportion of times mPATH-CheckIn is completed out of the total times mPATH-CheckIn should have been handed out; usage is calculated for nurses/providers as the proportion of times mPATH-CheckIn is completed and data is transmitted to the EHR out of the total times mPATH-CheckIn should have been handed out
Time Frame: up to month 6
Reporting Status: Not Posted

6. Secondary Outcome: mPATH-CRC Implementation Fidelity
Description: The proportion of patients who use mPATH-CRC and request a CRC screening test who have a test ordered or have the order dismissed (i.e., "self-order" feature is used as designed) in months 1-6
Time Frame: up to month 6
Reporting Status: Not Posted

7. Secondary Outcome: mPATH-CRC Maintenance
Description: The proportion of patients aged 50-74 who are eligible for CRC screening who complete mPATH-CRC or have risk factors identified by mPATH-CheckIn in months 7-12
Time Frame: months 7-12
Reporting Status: Not Posted

8. Secondary Outcome: mPATH-CheckIn Maintenance
Description: The proportion of patients aged 18 or older who complete mPATH-CheckIn in months 7-12
Time Frame: months 7-12
Reporting Status: Not Posted

9. Secondary Outcome: CRC Screening Tests Ordered
Description: The outcome is defined as the proportion of patients aged 50-74 who are eligible for CRC screening who have a CRC screening test ordered (colonoscopy, flexible sigmoidoscopy, fecal testing for blood, or fecal DNA testing) within 16 weeks of their index visit to the clinic. This outcome will also be compared between the pre- and post-implementation cohorts.
Time Frame: up to 16 weeks from index visit
Reporting Status: Not Posted

10. Secondary Outcome: mPATH-CRC Effectiveness
Description: The proportion of patients aged 50-74 who are eligible for CRC screening who complete CRC screening within 16 weeks of their index visit to the clinic. Effectiveness is determined by comparing the proportion who complete screening in a pre-implementation cohort (months 12 - 4 before implementation) to a post-implementation cohort (months 1 - 8 after implementation).
Time Frame: up to 16 weeks from index visit
Reporting Status: Not Posted

11. Secondary Outcome: Facilitators and Barriers to Maintenance (Sustained Use of mPATH-CRC Over Time)
Description: These will be identified through semi-structured interviews. Interviews will explore how mPATH-CRC was incorporated in the clinic's work flow and factors that affected maintenance such as intervention adaptations, organizational characteristics, and the champion's role. Interviews will be conducted with four members of each selected clinic: the clinic champion, one clinician, one front desk team member, and one medical assistant/nursing team member.
Time Frame: Month 12 or month of discontinuation of mPATH use
Reporting Status: Not Posted

12. Secondary Outcome: mPATH-CRC Reach (by Month)
Description: The proportion of patients aged 50-74 who are eligible for CRC screening who complete mPATH-CRC or have risk factors identified by mPATH-CheckIn in months 1-5 following implementation
Time Frame: Months 1-5
Reporting Status: Not Posted

13. Secondary Outcome: mPATH-CRC Acceptability
Description: The Acceptability of Intervention Measure (AIM) is a 4-item measure scored on a 5-point scale and summed. The Range of Scores is from 4 to 20. Higher Scores indicate higher acceptability.
Time Frame: month 6
Reporting Status: Not Posted

14. Secondary Outcome: mPATH-CRC Appropriateness
Description: The Intervention Appropriateness Measure (IAM) is a 4-item measure scored on a 5-point scale and summed. The Range of Scores is from 4 to 20. Higher Scores indicate higher appropriateness.
Time Frame: month 6
Reporting Status: Not Posted

15. Secondary Outcome: mPATH-CRC Feasibility
Description: The Feasibility of Intervention Measure (FIM) is a 4-item measure scored on a 5-point scale and summed. The Range of Scores is from 4 to 20. Higher Scores indicate higher feasibility.
Time Frame: month 6
Reporting Status: Not Posted

16. Secondary Outcome: mPATH-CheckIn Acceptability
Description: as for outcome 13
Time Frame: month 6
Reporting Status: Not Posted

17. Secondary Outcome: mPATH-CheckIn Appropriateness
Description: as for outcome 14
Time Frame: month 6
Reporting Status: Not Posted

18. Secondary Outcome: mPATH-CheckIn Feasibility
Description: as for outcome 15
Time Frame: month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Post-Implementation): English or Spanish-speaking patients aged 50-74 who are eligible for CRC screening who are seen in the study clinics randomized to mPATH utilizing the "low touch" implementation strategy in the 12 months after implementation.
  mPATH-CRC: mPATH-CRC is a self-administered iPad program that patients eligible for CRC screening use in primary care clinics to help them receive CRC screening.
  mPATH-Checkin: The mPATH-CheckIn program includes health questions to assist clinics with patient check-in, thereby incentivizing its use for all patients.
  "low touch" Implementation Strategy: Clinics randomized to receive the low touch implementation strategy will receive: Pre-Implementation Activities
  • N/A
  Implementation Kick-Off (Day 1)
  • On-site training with key clinic personnel
  Months 1 - 6
  * Phone/email technical support, as needed.
  * Access to web-based QA dashboard
  Months 7 - 12
  * Phone/email technical support, as needed
  * Access to web-based QA dashboard
Arm/Group | Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Post-Implementation) | Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Post-Implementation) | All Adult Clinic Patients on "High Touch" Strategy (Post-Implementation) | All Adult Clinic Patients on "Low Touch" Strategy (Post-Implementation) | Clinic Personnel on "High Touch" Strategy (Post-Implementation) | Clinic Personnel on "Low Touch" Strategy (Post-Implementation) | Clinic Patients Eligible for CRC Screening on "High Touch" Strategy (Pre-Implementation) | Clinic Patients Eligible for CRC Screening on "Low Touch" Strategy (Pre-Implementation)
All-Cause Mortality (participants affected / at risk) | 0/7933 | 0/5159 | 0/43775 | 0/23359 | 0/282 | 0/232 | 0/5526 | 0/3971
Serious Adverse Events (participants affected / at risk) | 0/7933 | 0/5159 | 0/43775 | 0/23359 | 0/282 | 0/232 | 0/5526 | 0/3971
Other Adverse Events (participants affected / at risk) | 0/7933 | 0/5159 | 0/43775 | 0/23359 | 0/282 | 0/232 | 0/5526 | 0/3971

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03843957/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT03843957/ICF_001.pdf